CLINICAL TRIAL: NCT07066995
Title: Dual-Target Chimeric Antigen Receptor (CAR) T-Cell Therapy Directed Against Mesothelin and Claudin 18.2 in Patients With Advanced or Metastatic Pancreatic Cancer
Brief Title: Mesothelin and Claudin 18.2 Dual-Target CAR-T Therapy in Advanced Pancreatic Cancer
Acronym: BAH2573-102
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202571-102
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer; Pancreatic Carcinoma; Pancreatic Cancer Non-resectable; Pancreatic Cancer Stage IV
Keywords: Pancreatic Cancer; claudin 18.2; Pancreatic Carcinoma; CAR-T; Mesothelin
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Mesothelin

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2, first-in-human, open-label, non-randomized trial of sequential dual-target CAR-T cell therapy in subjects with advanced pancreatic cancer
Masking Description: Open-label clinical trials are a category of clinical research where the masking is minimal or nonexistent. In such trials, both the participants and the researchers are fully aware of the treatment assignments, which means participants know the treatment they are receiving, and researchers are aware of each participant's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesothelin and Claudin 18.2 CAR T cells, chemotherapy (Experimental): Patients will be administered fludarabine phosphate intravenously (IV) over a 30-minute period on days -4 to -2. Additionally, cyclophosphamide will be administered intravenously (IV) over 60 minutes on day -2. Subsequently, patients will receive Mesothelin and Claudin 18.2 CAR T cells intravenously (IV) over a duration of 10-20 minutes on day 0. Patients who exhibit positive responses to the initial dose of Mesothelin and Claudin 18.2 CAR T cells, do not experience unacceptable side effects, and have a sufficient quantity of cells available may be eligible to receive 2 or 3 additional doses of Mesothelin and Claudin 18.2 CAR T cells.
  Interventions: Biological: Mesothelin and Claudin 18.2 CAR-T cells

INTERVENTIONS:
Biological: Mesothelin and Claudin 18.2 CAR-T cells — The intervention in this clinical trial involves a novel approach using Mesothelin and Claudin 18.2 Chimeric Antigen Receptor T (CAR T) cells combined with chemotherapy. The goal is to assess safety and efficacy in patients with specific hematologic malignancies.
  Treatment Regimen:
  Fludarabine Phosphate (Days -4 to -2): IV administration of fludarabine phosphate over 30 minutes on days -4 to -2. It's part of the preparatory regimen to enhance the body's response to CAR T-cell therapy.
  Cyclophosphamide (Day -2): IV cyclophosphamide over 60 minutes on day -2.
  Mesothelin and Claudin 18.2 Chimeric Antigen Receptor T Cells (Day 0): IV administration of investigational therapy, Mesothelin and Claudin 18.2 CAR T cells, over 10-20 minutes on day 0.
  Additional Doses: Eligible patients responding well to the initial Mesothelin and Claudin 18.2 CAR-T cell infusion without unacceptable side effects and sufficient CAR-T cell availability may receive 2 or 3 additional doses.

SUMMARY:
Autologous T-cells engineered to express CARs targeting Mesothelin and Claudin18.2, for Unresectable locally advanced or metastatic pancreatic adenocarcinoma (Pancreatic Ductal Adenocarcinoma, PDAC), administered as two separate sequential infusions following lymphodepleting chemotherapy

DETAILED DESCRIPTION:
Pancreatic cancer is one of the most lethal malignancies, with a poor prognosis in advanced stages. Mesothelin (MSLN) and Claudin 18.2 (CLDN18.2) are tumor-associated antigens overexpressed in pancreatic adenocarcinoma cells. Both are promising immunotherapy targets, as they are prevalent in pancreatic tumors while largely restricted in normal tissues. CAR-T cell therapies directed at these antigens have shown early evidence of safety and anti-tumor activity. For example, mesothelin-specific CAR T cells have achieved stable disease and metabolic tumor regression in initial trials without dose-limiting toxicity. Similarly, CLDN18.2-specific CAR-T cells yielded objective remissions (including complete remission) in refractory pancreatic cancer, albeit with some gastric mucosal toxicity due to low-level target expression in normal stomach. Targeting two antigens may improve tumor control by addressing antigen heterogeneity and reducing immune escape. This trial evaluates a dual-target CAR-T strategy, in which two separate CAR-T products (one for mesothelin, one for claudin18.2) are given sequentially.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival time ≥3 months;
* Histologically or cytologically confirmed pancreatic adenocarcinoma that is advanced (unresectable or metastatic). Patients should have received, or be intolerant of, standard first-line therapy (e.g., gemcitabine/nab-paclitaxel, FOLFIRINOX) for advanced disease. A short course of current first-line therapy is allowed for the purpose of bridging to manufacturing, but evidence of disease progression on or after at least one line is required prior to infusion (for the dose-expansion phase, patients must have progressed on ≥1 prior systemic regimen).
* ECOG Performance Status: 0 or 1 (fully active or restricted in strenuous activity but ambulatory).
* Liver and kidney function, cardiopulmonary function meet the following requirements:
* Creatinine ≤1.5×ULN; (2) Electrocardiogram showed no clinically significant abnormal bands;
* Blood oxygen saturation >91% in non-oxygen state;
* Total bilirubin ≤2×ULN; ALT and AST≤2.5 x ULN; ALT and AST abnormalities due to disease, such as liver infiltration or bile duct obstruction, were determined to be less than 5×ULN. If Gilbert syndrome is diagnosed, the total bilirubin index can be relaxed to ≤3.0×ULN and the direct bilirubin ≤1.5×ULN.
* No serious mental disorders;
* Can understand this test and has signed the informed consent.

Exclusion Criteria:

* Hepatitis B surface antigen (HBsAg) positive; Hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal reference value range; Hepatitis C virus (HCV) Antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; Human immunodeficiency virus (HIV) Antibody positive; Syphilis positive;
* Serious heart disease, including but not limited to unstable angina, myocardial infarction or bypass or stent surgery (within 6 months prior to screening), congestive heart failure (NYHA classification ≥III), and severe arrhythmia;
* Systemic diseases that are deemed unstable by researchers: including but not limited to severe liver, kidney, or metabolic diseases that require drug treatment;
* Active or uncontrollable infections (except mild genitourinary and upper respiratory tract infections) that require systemic treatment within 7 days prior to administration;
* Pregnant or lactating women, and female subjects who plan pregnancy within 2 years after cell transfusion or male subjects whose partners plan pregnancy within 2 years after cell transfusion;
* Patients who received CAR-T therapy or other gene-modified cell therapy before screening;
* Participated in other clinical studies 1 month before screening;
* Evidence of central nervous system invasion during subject screening;
* Mental patients with depression or suicidal thoughts;
* Situations considered unsuitable for inclusion by other researchers.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD19/BCMA chimeric antigen receptor (CAR) T cells | 28 days
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 at three dose levels until the maximum tolerated dose (MTD) is determined.

SECONDARY OUTCOMES:
Rate of successful manufacture and expansion of the Mesothelin and Claudin 18.2 chimeric antigen receptor (CAR) T cells | 60 days
  satisfy the targeted dose level and meet the required release specifications outlined in the Certificate of Analysis (COA)

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No